CLINICAL TRIAL: NCT04044599
Title: Lactobacillus for Luteal Phase Support to Improve IVF Outcomes
Brief Title: Lactobacillus for Luteal Phase Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Prof. Dr. Gürkan Uncu, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-11/24
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: IVF

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): THE GROUP THAT WİLL RECİEVE VAGİNAL LACTOBACİLLUS
  Interventions: Drug: Gynoflor
- Control (No Intervention): Control group

INTERVENTIONS:
Drug: Gynoflor — VAGİNAL GYNOFLOR
  Arms: Study

SUMMARY:
The aim of this study was to evaluate the effect of vaginal lactobacilli, a regulator of normal vaginal flora, on embryo implantation success during IVF / ICSI cycle follow-up.

DETAILED DESCRIPTION:
Urogenital region accounts for 9% of the total human microbiome. The role of vaginal microbioma in infertility and assisted reproductive technologies has not yet been clarified. It is thought that microorganisms such as mycoplasma, chlamydia and Neiseria gonorrhea are associated with infertility, and changes in subclinical microbiota such as bacterial vaginosis (BV) may be a risk factor for subfertility. The majority of the normal elements of the vaginal flora are the various Lactobacillus species. Lactobacilli constitute a healthy environment for the embryo in the pre- and peri-conception period. They are thought to support implantation not only by their presence but also by the lactic acid, hydrogen peroxide, bacteriocin and probiotics they produce. Bacterial vaginosis (BV) is the reduction of lactobacilli in the dominance of the vaginal microbiota and the transition of the microbial environment to the dominance of Gardnella vaginalis.The two main functions of lactobacilli in translating the balances in the reproductive system in favor of successful implantation and pregnancy rates; lactic acid production and H 2 O 2 recovery. It has been shown that up to 40% of patients undergoing in vitro fertilization (IVF) cycles have abnormal reproductive tract microbiata. To date, studies on vaginal microbiata and implantation have been carried out to identify vaginal microbiome by genetic sequencing of the vaginal specimens. In these studies, endometrial microbiota; When lactobacilli were classified as dominant (> 90%) and non-lactobacilli were dominant; In the presence of lactobacilli non-dominant microbiota, decreased implantation, pregnancy and ongoing pregnancy rates and more negative reproductive results were obtained.

To date, the limited number of studies evaluating the effects of lactobacilli on assisted reproductive methods success and implantation; vaginal or endometrial lactobacilli burden was evaluated. Therefore, for the first time in our study; The aim of this study was to evaluate the effect of vaginal lactobacilli, a regulator of normal vaginal flora, on embryo implantation success during IVF / ICSI cycle follow-up.The study group will be composed of patients who will receive 4 vaginal lactobacillus tablet immediately after the OPU procedure.The ones who will not receive vaginal lactobacillus tablets will compose the control group.

Patients will be selected from infertile patients that underwent IVF/ICSI protocol. There will be no change in the routine ovarian stimulation protocols and luteal phase support treatments that patients should receive routinely. Following ovulation induction with controlled ovarian stimulation (KOH), which is routinely administered in IVF treatment cycles, following the collection of oocytes, the luteal phase support is routinely recommended for the preparation of the endometrium to embryo transfer in artificial, stimulated cycles on the evening of the same day. If pregnancy occurs, luteal phase support should be continued for an average of 8 weeks. In fresh embryo transfer cycles, vaginal progesterone is routinely used for luteal phase support in all patients in our clinic. All patients will receive the same luteal phase treatment routinely.For the study the patients who will have day 5 good quality embryo transfer performed will be selected.

ELIGIBILITY:
Inclusion Criteria:

* having embryo transfer of a day 5 good quality embryo

Exclusion Criteria:

* Uterin pathologies
* Having additional adjuvants for luteal phase support
* Having day 3 embryo transfer

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-30 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 4 weeks after embryo transfer
  To see the gestational sac

SECONDARY OUTCOMES:
clinical pregnancy | 6 weeks after embryo transfer
  To see the fetal cardiac activity

OTHER OUTCOMES:
Ongoing pregnancy | 12 weeks after embryo transfer
  Ongoing pregnancy after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Uncu, Prof., Study Director — Uludag University
Locations (1):
- Uludag University ART Center, Bursa, Turkey (Türkiye)